CLINICAL TRIAL: NCT00739154
Title: Clinical Cohort Study of Association Between Steady State Phenytoin Treatment and Better Clinical Parameters of Glaucoma
Brief Title: Protective Effect of Phenytoin on Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: prof. Dov Weinberger, head of ophthalmology department, Rabin medical center
Other Study IDs: 005062; non
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Primary Open Angle Glaucoma; Secondary Open Angle Glaucoma; Narrow-Angle Glaucomas; Normal Tension Glaucoma
Keywords: glaucoma; Phenytoin; retinal nerve fiber layer; corrected pattern standard deviation; visual acuity; optic disc cupping
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Low Tension Glaucoma; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: glaucoma patients who also suffer from epileptic disorder and receiving chronic oral Phenytoin treatment
- 2: glaucoma patients who also suffer from epileptic disorder receiving anti-convulsant treatment other then Phenytoin
- 3: glaucoma patients with no epileptic disorder and not receiving anti-convulsant treatment

SUMMARY:
since glaucoma is considered an optic neuropathy, new treatments for glaucoma are being continuously investigated, including neuroprotection.

Previous studies implied that phenytoin, a potent anti-convulsive drug, has a neuroprotective role, and Na+ channels blockage was suggested as a possible mechanism.

This study predicts that glaucoma patients taking Phenytoin will have a less advanced glaucoma as compared to patients not taking the drug. Glaucoma severity will be determined by visual acuity, visual fields, optic disc cupping and nerve fiber layer thickness

DETAILED DESCRIPTION:
The study will examine adult patients who suffer from glaucoma and epileptic disorders on the same time. the study group will include glaucoma patients, being treated with oral Phenytoin for their epileptic disorder. The study group will be compared to 2 control groups:

* Glaucoma patients with epileptic disorder,receiving different medication than Phenytoin
* Glaucoma patients with no epileptic disorder.

  4 parameters will be evaluated for all groups:
  1. Best corrected visual acuity
  2. Optic disc cupping
  3. visual fields and general perimetric indices
  4. peripapillary retinal nerve fiber layer.

Every participant in the study,after giving his informed consent, will be evaluated by a senior ophthalmologist in a single office appointment. The appointment will include a visual acuity, complete ophthalmic examination,Humphrey perimetric visual field testing and peripapillary RNFL thickness measurement by OCT.

no drug or other treatment will be given to the participants

after data collection, average +/-Standard deviation for the 4 parameters will be compared between the 3 groups. Student T-test and one- way ANOVA will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of glaucoma
* chronic treatment with phenytoin for any indication

Exclusion Criteria:

* pregnancy
* visual acuity less then 6/60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of a tertiary hospital's specialized epilepsy clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
peripapillary RNFL thickness | immediate

SECONDARY OUTCOMES:
corrected pattern standard deviation in perimetric visual field | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Omer Y Bialer, MD, Study Director — Rabin medical center, Petah Tikva, Israel; Dan Gaa'ton, MD, Study Director — Rabin medical center, Petah-Tikva, Israel
Locations (1):
- Beilinson hospital, Rabin medical center, Petah Tikva, Israel

REFERENCES:
- [Background] Chidlow G, Wood JP, Casson RJ. Pharmacological neuroprotection for glaucoma. Drugs. 2007;67(5):725-59. doi: 10.2165/00003495-200767050-00006. PMID 17385943
- [Background] Ben Simon GJ, Bakalash S, Aloni E, Rosner M. A rat model for acute rise in intraocular pressure: immune modulation as a therapeutic strategy. Am J Ophthalmol. 2006 Jun;141(6):1105-11. doi: 10.1016/j.ajo.2006.01.073. PMID 16765680
- [Background] Willmore LJ. Antiepileptic drugs and neuroprotection: current status and future roles. Epilepsy Behav. 2005 Dec;7 Suppl 3:S25-8. doi: 10.1016/j.yebeh.2005.08.006. Epub 2005 Oct 18. PMID 16239127
- [Background] Huang D, Swanson EA, Lin CP, Schuman JS, Stinson WG, Chang W, Hee MR, Flotte T, Gregory K, Puliafito CA, et al. Optical coherence tomography. Science. 1991 Nov 22;254(5035):1178-81. doi: 10.1126/science.1957169.
- [Background] Mills RP, Budenz DL, Lee PP, Noecker RJ, Walt JG, Siegartel LR, Evans SJ, Doyle JJ. Categorizing the stage of glaucoma from pre-diagnosis to end-stage disease. Am J Ophthalmol. 2006 Jan;141(1):24-30. doi: 10.1016/j.ajo.2005.07.044. PMID 16386972
- [Result] Klein BE, Klein R, Sponsel WE, Franke T, Cantor LB, Martone J, Menage MJ. Prevalence of glaucoma. The Beaver Dam Eye Study. Ophthalmology. 1992 Oct;99(10):1499-504. doi: 10.1016/s0161-6420(92)31774-9. PMID 1454314
- [Result] Ates O, Cayli SR, Gurses I, Turkoz Y, Tarim O, Cakir CO, Kocak A. Comparative neuroprotective effect of sodium channel blockers after experimental spinal cord injury. J Clin Neurosci. 2007 Jul;14(7):658-65. doi: 10.1016/j.jocn.2006.03.023. PMID 17532502
- [Result] Podos SM, Becker B, Beaty C, Cooper DG. Diphenylhydantoin and cortisol metabolism in glaucoma. Am J Ophthalmol. 1972 Sep;74(3):498-500. doi: 10.1016/0002-9394(72)90915-4. No abstract available. PMID 5053695
- [Result] Naskar R, Quinto K, Romann I, Schuettauf F, Zurakowski D. Phenytoin blocks retinal ganglion cell death after partial optic nerve crush. Exp Eye Res. 2002 Jun;74(6):747-52. doi: 10.1006/exer.2002.1173. PMID 12126947
- [Result] Lo AC, Black JA, Waxman SG. Neuroprotection of axons with phenytoin in experimental allergic encephalomyelitis. Neuroreport. 2002 Oct 28;13(15):1909-12. doi: 10.1097/00001756-200210280-00015. PMID 12395089
- [Result] Hains BC, Waxman SG. Neuroprotection by sodium channel blockade with phenytoin in an experimental model of glaucoma. Invest Ophthalmol Vis Sci. 2005 Nov;46(11):4164-9. doi: 10.1167/iovs.05-0618. PMID 16249495
- [Result] Savini G, Bellusci C, Carbonelli M, Zanini M, Carelli V, Sadun AA, Barboni P. Detection and quantification of retinal nerve fiber layer thickness in optic disc edema using stratus OCT. Arch Ophthalmol. 2006 Aug;124(8):1111-7. doi: 10.1001/archopht.124.8.1111. PMID 16908813
- [Result] Carpineto P, Ciancaglini M, Zuppardi E, Falconio G, Doronzo E, Mastropasqua L. Reliability of nerve fiber layer thickness measurements using optical coherence tomography in normal and glaucomatous eyes. Ophthalmology. 2003 Jan;110(1):190-5. doi: 10.1016/s0161-6420(02)01296-4. PMID 12511365
- [Result] Williams ZY, Schuman JS, Gamell L, Nemi A, Hertzmark E, Fujimoto JG, Mattox C, Simpson J, Wollstein G. Optical coherence tomography measurement of nerve fiber layer thickness and the likelihood of a visual field defect. Am J Ophthalmol. 2002 Oct;134(4):538-46. doi: 10.1016/s0002-9394(02)01683-5. PMID 12383810
- [Result] Budenz DL, Chang RT, Huang X, Knighton RW, Tielsch JM. Reproducibility of retinal nerve fiber thickness measurements using the stratus OCT in normal and glaucomatous eyes. Invest Ophthalmol Vis Sci. 2005 Jul;46(7):2440-3. doi: 10.1167/iovs.04-1174. PMID 15980233
- [Result] Leung CK, Chan WM, Chong KK, Yung WH, Tang KT, Woo J, Chan WM, Tse KK. Comparative study of retinal nerve fiber layer measurement by StratusOCT and GDx VCC, I: correlation analysis in glaucoma. Invest Ophthalmol Vis Sci. 2005 Sep;46(9):3214-20. doi: 10.1167/iovs.05-0294. PMID 16123421